CLINICAL TRIAL: NCT00972153
Title: Reduction of Airborne Particulate in the Surgical Field Using Directed Local Airflow
Brief Title: Device to Reduce Surgery Site Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nimbic Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ABS001-0912403
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Results first posted 2010-05-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Surgery
Keywords: Decrease in CFU density at surgery site; Decrease in airborne particulate at surgery site

ARMS (3):
- No device used (No Intervention)
- Device attached, not activated (Sham Comparator)
  Interventions: Device: Sham Air Barrier System device
- Device deployed and activated (Experimental)
  Interventions: Device: Air Barrier System Device

INTERVENTIONS:
Device: Air Barrier System Device — Device is deployed adjacent to the surgery site and activated so that the filtered air emits over the surgery site.
  Arms: Device deployed and activated
Device: Sham Air Barrier System device — Device is deployed to the surgery site, but the airflow is not activated. This intervention is used to determine any effects that the presence of the device alone may have.
  Arms: Device attached, not activated

SUMMARY:
The objective of this study is to determine whether the Air Barrier System device reduces airborne particulate and airborne colony forming units present at a surgery site.

DETAILED DESCRIPTION:
The Air Barrier System is a device that uses localized clean air flow to shield a surgery site from ambient airborne contamination. This study examines the hypothesis that the Air Barrier System can reduce the presence of airborne colony-forming units (e.g. bacteria colonies) and particulate at the surgery site.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for primary total hip arthroplasty

Exclusion Criteria:

* Prior history of infection
* Revision arthroplasty
* Screens positive for MRSA
* Undergoing hemiarthroplasty or resurfacing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Stocks, MD, Principal Investigator — Fondren Orthopaedic Group
Locations (1):
- Texas Orthopedic Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Stocks GW, Self SD, Thompson B, Adame XA, O'Connor DP. Predicting bacterial populations based on airborne particulates: a study performed in nonlaminar flow operating rooms during joint arthroplasty surgery. Am J Infect Control. 2010 Apr;38(3):199-204. doi: 10.1016/j.ajic.2009.07.006. Epub 2009 Nov 12. PMID 19913327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six patients of the surgeon who consented to undergo primary total hip arthroplasty between May and September 2009 were recruited to participate in this study. All consenting patients were eligible. Patients undergoing hemiarthroplasty, resurfacing, or revision arthroplasty were excluded from recruitment.
Period: Overall Study
Arm/Group | No Device Used | Device Attached, Not Activated | Device Deployed and Activated
Started | 12 | 12 | 12
Completed | 12 | 11 (One case excluded due to technical problem with measuring equipment.) | 12
Not Completed | 0 | 1 | 0
Not completed — Equipment malfunction during case | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Device Used | Device Attached, Not Activated | Device Deployed and Activated | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 8 | 25
  >=65 years | 4 | 3 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 20
  Male | 5 | 6 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Surgery Site CFU Density
Description: Colony forming unit counts were collected from the air within 5 cm of the surgical wound using a bioaerosol "slit" sampling device. Air was drawn through a sterile PVC tubing located at the incision and impacted upon media (TSA 5% sheep's blood) plates located in the sampling device. The plates were exchanged every 10 minutes throughout the procedure. Values are presented as CFU/cubic meter.
Time Frame: Ten minute intervals throughout surgery
Population: Airborne CFU densities were obtained in ten-minute intervals throughout each procedure. Average surgery duration was 69 minutes in the control and sham groups; 66 minutes in the experiment group. A total of 208 density readings were obtained.
Measure: Median (Full Range); unit: CFU/cubic meter
Arm/Group | No Device Used | Device Attached, Not Activated | Device Deployed and Activated
Number analyzed (Participants) | 12 | 11 | 12
CFU/cubic meter | 7 [0 to 36] | 11 [0 to 46] | 0 [0 to 14]
Statistical Analysis 1: Comparison: No Device Used vs Device Attached, Not Activated vs Device Deployed and Activated; Descriptive statistics (means, medians, frequencies) were used to evaluate the distributions of variables. One-way analysis of variance and independent t-tests or Mann-Whitney U tests were used to compare patient and environmental characteristics between groups. Generalized estimating equations were used to evaluate the effects of group and other factors on airborne CFUs/cubic meter at the surgical site in each 10 minute interval; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Surgery Site Particulate Density (Size >10 Micrometer)Per Cubic Meter
Description: Airborne particulate was measured using a particle analyzer (LASAIR II 310B). The analyzer sampled continuously during surgery at a rate of 28.3 L/min and recorded data at one-minute intervals. The samples were collected through a length of sterile PVC tubing with the end placed adjacent to the CFU sample tubing, within 5 cm of the surgical incision. Particles of various diameters were obtained; particles of size >10 micrometer had the strongest correlation to the presence of CFUs at the incision site.
Time Frame: Ten minute intervals throughout surgery
Measure: Median (Full Range); unit: >10 micrometer particles / cubic meter
Arm/Group | No Device Used | Device Attached, Not Activated | Device Deployed and Activated
Number analyzed (Participants) | 12 | 11 | 12
>10 micrometer particles / cubic meter | 1377 [459 to 8746] | 1165 [424 to 5474] | 247 [0 to 5968]
Statistical Analysis 1: Comparison: No Device Used vs Device Attached, Not Activated vs Device Deployed and Activated; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | No Device Used | Device Attached, Not Activated | Device Deployed and Activated
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No